CLINICAL TRIAL: NCT04112472
Title: Clinical Trial - ES 900 - 2019
Brief Title: Clinical Trial ES 900 - 2019
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haag-Streit AG (Industry)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1023551
Record Dates: First submitted 2019-09-20; First posted 2019-10-02 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Optical Biometry of the Human Eye; General Analysis of the Anterior Chamber of the Human Eye

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Examination of participants (Experimental): Examination of participants by means of the investigational device as well as the comparative devices.
  Interventions: Device: EYESTAR 900

INTERVENTIONS:
Device: EYESTAR 900 — EYESTAR 900 is an optical biometry device used to create a geometrical representation of the eye by means of optical interferometry. The intervention are optical, non-contact examinations with the investigational device EYESTAR 900 and comparative device(s). Results of the examinations serve to compare the performance data of the investigational device with those of the comparative devices.

SUMMARY:
The primary objective of this clinical trial is to assess the clinical performance of the investigational device. To that end, the Limits of Agreement with respect to comparator devices are analyzed. The Limits of Agreement allow estimating the expected measurement deviation per measurand, which is compared to the "maximum acceptable measurement error", as defined by the Risk Analysis of the investigational device, to assess the risk involved in measurements of the investigational device. Furthermore, the in-vivo repeatability will be quantified for each measurand, as well as the confidence intervals for mean deviation with respect to the current gold standard device.

As a secondary objective of the study, raw measurement data will be collected to allow for improvement of existing algorithms, development of additional measurands and for retrospective analysis.

DETAILED DESCRIPTION:
The EYESTAR900 (the investigational device) is a new device by HAAG-STREIT AG, for measurement of optical biometry and advanced corneal topography by swept-source optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

At least one eye of each subject needs to fulfill one of the following inclusion criteria:

* volunteers with normal phakic eye;
* patients seeking cataract surgery;
* patients with pseudophakic eye;
* patients with oil-filled eye;
* patients with aphakic eye.

Exclusion Criteria:

* Exclusion criteria per subject:

  * underage patients (younger than 18 years);
  * vulnerable patients;
  * inability to give informed consent;
* Exclusion criteria per eye:

  * inability to maintain stable fixation;
  * corneal lesions or scarring;
  * previous corneal surgery (except: pseudophakic eyes, oil-filled eyes, aphakic eyes);
  * previous intraocular surgery (except: pseudophakic eyes, oil-filled eyes, aphakic eyes);
  * active inflammation of the eye;
  * active infection of the eye;
  * tear film break up time of less than 5 sec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Keratometry Measurand: Kmean (Spherical refractive power of central cornea) in keratometric diopters [dpt] | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator device for Kmean.
Keratometry Measurand: AST (Anterior central corneal astigmatism) in [dpt] | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator device for AST.
Keratometry Measurand: Axis (Anterior steep meridian angle) in [°] | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator device for Axis. Axis is the angle of the anterior central corneal astigmatism.
  The value of Axis is measured in [°], whereas the differences shall be expressed in [dpt].
Axial Measurand: AL (Axial length) in [mm] | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator device for AL. AL is measured from the corneal tear film to the inner limiting membrane.
Axial Measurand: CCT (Corneal thickness) in [μm] | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator device for CCT. CCT is measured from the corneal tear film to the corneal endothelium.
Axial Measurand: ACD (Anterior chamber depth) in [mm] | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator device for ACD. ACD is measured from the corneal tear film to the anterior surface of the lens.
Axial Measurand: LT (Lens thickness) in [mm] | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator device for LT. LT is measured from the anterior to the posterior surface of the lens.
Imaging Measurand: WTW (White-to-White) in [mm] | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator devices for WTW. WTW distance is the horizontal diameter of a best fit circle to the iris border.
Imaging Measurand: ICX / ICY (Iris barycenter in horizontal direction / in vertical direction) in [mm] | Through study completion, approximately 7 months.
  In-vivo repeatability of investigational and comparator device for Iris barycenter. The iris barycenter is the displacement of the iris center relative to the vertex in X (horizontal direction) and Y (vertical direction) coordinates.
Imaging Measurand: PD (Pupil diameter) in [mm] | Through study completion, approximately 7 months.
  In-vivo repeatability of investigational and comparator device for PD. PD is measured at the diameter of a best fit circle to the pupil border.
Imaging Measurand: PCX / PCY (Pupil barycenter in horizontal direction / in vertical direction) in [mm] | Through study completion, approximately 7 months.
  In-vivo repeatability of investigational and comparator device for Iris barycenter. The pupil barycenter is the displacement of the iris center relative to the vertex in X (horizontal direction) and Y (vertical direction) coordinates.
Anterior corneal topography: Elevation (Anterior torical elevation) in [µm] (2D-map) | Through study completion, approximately 7 months.
  In-vivo repeatability and confidence interval of mean deviation with respect to comparator device, for elevation in [µ]; axial curvature in [dpt].
Anterior corneal topography: Axial curvature (Anterior tangential curvature) in [dpt] (2D-map) | Through study completion, approximately 7 months.
  In-vivo repeatability and confidence interval of difference between investigational and comparator devices for Anterior torical elevation. The measuring performance over the 2D-map is subdivided in three zones (central zone, middle zone, peripheral zone).
Posterior corneal topography: Elevation (Posterior torical elevation) in [µm] (2D-map) | Through study completion, approximately 7 months.
  In-vivo repeatability of investigational and comparator device for Posterior torical elevation. The measuring performance over the 2D-map is subdivided in three zones (central zone, middle zone, peripheral zone).
Posterior corneal topography: Axial curvature (Posterior tangential curvature) in [dpt] (2D-map) | Through study completion, approximately 7 months.
  In-vivo repeatability and confidence interval of differences of investigational and comparator devices for Posterior tangential curvature. The measuring performance over the 2D-map is subdivided in three zones (central zone, middle zone, peripheral zone).
Corneal pachymetry: Corneal thickness map in [µm] | Through study completion, approximately 7 months.
  In-vivo repeatability and confidence interval of differences of investigational and comparator device for Corneal thickness map. The measuring performance over the 2D-map is subdivided in three zones (central zone, middle zone, peripheral zone).
Simulated Keratometry: SimKmean (Mean simulated keratometry) in [dpt] | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator devices for SimKmean.
Simulated Keratometry: SimAST (Simulated astigmatism) in [dpt] | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator devices for SimAST.
Simulated Keratometry: SimAxis (Simulated keratometry anterior steep meridian angle) in [°] | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator device for SimAxis. The value of Axis is measured in [°], whereas the differences shall be expressed in [dpt]. SimAxis is the angle of the larger simulated keratometry radius with respect to the horizontal axis X.
Simulated Keratometry: Anterior corneal shape factor (E): Dimensionless quantity | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator device for Anterior corneal shape factor (E), that characterizes the anterior corneal asphericity.
Simulated Posterior Keratometry: SimPKmean (Mean simulated posterior keratometry) in [dpt] | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator device for SimPKmean. SimPKmean is the corresponding refractive power in diopters.
Simulated Posterior Keratometry: SimPAST (Simulated keratometry posterior corneal astigmatism) in [dpt] | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator device for SimPAST.
Simulated Posterior Keratometry: SimPAxis (Simulated keratometry posterior steep meridian angle) in [°] | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator device for SimPAxis. SimPAxis represents the angle of the larger simulated keratometry radius of curvature with respect to the horizontal axis X.
Simulated Posterior Keratometry: Posterior corneal shape factor (PE): Dimensionless quantity | Through study completion, approximately 7 months.
  In-vivo repeatability, limits of agreement and confidence interval of difference between investigational and comparator device for Posterior corneal shape factor (PE), that characterizes the posterior corneal asphericity.

OTHER OUTCOMES:
Acquisition of volumetric OCT Data of the eye. | Through study completion, approximately 7 months
  The data is collected to allow for: Improvement of existing algorithms, development of additional measurands and for retrospective analysis. The data will not be processed within the scope of this clinical trial.
Acquisition of photographic images of the eye. | Through study completion, approximately 7 months
  The data is collected to allow for: Improvement of existing algorithms, development of additional measurands and for retrospective analysis. The data will not be processed within the scope of this clinical trial.

CONTACTS AND LOCATIONS:
Overall Officials: David Goldblum, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hopital Basel, Basel, Switzerland